CLINICAL TRIAL: NCT02166944
Title: The Study of Tamoxifen Treatment in Patients With Motor Neuron Disease
Brief Title: Tamoxifen Treatment in Patients With Motor Neuron Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201307022
Record Dates: First submitted 2014-06-09; First posted 2014-06-18 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2014-06

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS Functional Ration Scale; TAR-DNA-binding Protein-43; Tamoxifen; mTOR
Keywords: amyotrophic lateral sclerosis; ALS functional ration scale; TAR-DNA-binding protein-43; tamoxifen; mTOR
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tamoxifen (Experimental): tamoxifen 40 mg daily for one year
  Interventions: Drug: tamoxifen 40 mg daily for one year
- placebo (Placebo Comparator): placebo drugs
  Interventions: Drug: tamoxifen 40 mg daily for one year

INTERVENTIONS:
Drug: tamoxifen 40 mg daily for one year — both arms with riluzole daily
  Other Names: Nolvadex

SUMMARY:
The aim of this study is to survey the effect of Tamoxifen in motor neuron disease (MND) patients, amyotrophic lateral sclerosis (ALS) with regular riluzole usage. TDP-43 is related to ALS. Increased the ubiquitinated or phosphorylated TDP-43 can cause animal model of ALS, and TDP43 can be degraded either by proteasome or autophagy pathway system. Autophagy pathway can be activated by mTOR inhibition, resulting in ameliorating TDP-43 accumulation and rescue in motor function in animal model. Tamoxifen had shown ability of enhance both proteasome and autophagy pathway, therefore the investigators assume that Tamoxifen probably can ameliorate TDP-43 accumulation and inclusion body formation in ALS.

DETAILED DESCRIPTION:
The investigators will assess the ALSFR-s in ALS patients at start, 1, 3, 6 and 12 months and correlate the score to the neurological outcome of the patients with and without tamoxifen treatment at dose of 40mg daily for one year.

The study will be able to prove the investigators hypothesis: Tamoxifen, a protease and autophagy enhancer, has synergic effect with riluzole in ALS patients to slowing the progression of neurological dysfunction, and respiratory insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed and confirmed ALS patients, with regular follow up and oral form riluzole at National Taiwan University or Shuang- Ho Hospital for more than 6 months.
2. Age ≧20 years old

Exclusion Criteria:

1. Patients who had already ventilator dependent, not regular followed up for more than 6 months or against medical advice, refuse to follow up at neurology department will be excluded in this study.
2. Patients with now or previous usage of Tamoxifen
3. Patients with any contraindications of Tamoxifen usage
4. Patients with other internal medicine illiness

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Amyotrophic Lateral Sclerosis Functional Ration Scales (ALSFRS) at 1, 3, 6,12 months | Baseline, month 1, 3, 6, 12
  Amyotrophic Lateral Sclerosis Functional Ration Scales (ALSFRS) measured by a neurologist

SECONDARY OUTCOMES:
Change from Baseline in pulmonary function test at 1, 3, 6,12 months | baseline, month 1, 3, 6, 12
  Expiratory reserve volume (ERV) Forced vital capacity (FVC) Forced expiratory volume (FEV) Forced expiratory flow 25% to 75% Functional residual capacity (FRC) Maximum voluntary ventilation (MVV)
  * Residual volume (RV)
  * Peak expiratory flow (PEF).
  * Slow vital capacity (SVC)
  * Total lung capacity (TLC)

OTHER OUTCOMES:
Change from Baseline in blood TDP43 related biomarkers at 1, 3, 6,12 months | baseline, month 1, 3, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Chaur-Jong Hu, M.D., Principal Investigator — Shung Ho Hospital, Taipei Meidcal University
Locations (1):
- Po-Chih Chen, New Taipei City, Taiwan

REFERENCES:
- [Derived] Trist BG, Fifita JA, Hogan A, Grima N, Smith B, Troakes C, Vance C, Shaw C, Al-Sarraj S, Blair IP, Double KL. Co-deposition of SOD1, TDP-43 and p62 proteinopathies in ALS: evidence for multifaceted pathways underlying neurodegeneration. Acta Neuropathol Commun. 2022 Aug 25;10(1):122. doi: 10.1186/s40478-022-01421-9. PMID 36008843